CLINICAL TRIAL: NCT03716271
Title: The Light Sword Lens - a Novel Method of Presbyopia Compensation: a Pilot Clinical Study
Brief Title: The Light Sword Lens for Presbyopia Compensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Collaborators: Warsaw University of Technology (Other)
Responsible Party: Principal Investigator, Marek Rekas, Professor, Military Institute od Medicine National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSL
Record Dates: First submitted 2018-10-10; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Presbyopia
Keywords: presbyopia compensation; EDF; Light Sword Lens
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Visual Acuity Examination with a novel lens — Visual Acuity Examination with a novel lens set in an ophthalmic trial frame

SUMMARY:
Clinical assessment of a new optical element for presbyopia compensation - the Light Sword Lens.

DETAILED DESCRIPTION:
Healthy dominant eyes of presbyopes were examined for visual performance. The examination was performed in the ophthalmic trial frame, which included assessment of 3 trials: reference (with lens for distance correction); stenopeic (distance correction with a pinhole ϕ=1,25 mm) and Light Sword Lens (distance correction with a Light Sword Lens). In each trial, visual acuity was assessed in 7 tasks for defocus from 0.2D to 3.0D while contrast sensitivity in 2 tasks for defocus 0.3D and 2.5D.

ELIGIBILITY:
Inclusion Criteria:

* emmetropic or hyperopic eyes with a spherical error of maximum +1.75D and astigmatism of ≤ 0.5D.
* Corrected distance visual acuity (CDVA) had to be better than 0.1 logMAR (20/25) and at the same time contrast sensitivity (CS) could not be less than 1.9 logCS. -Uncorrected near visual acuity was required to be worse than 0.4 logMAR (20/50), as a proof of presbyopia.

Exclusion Criteria:

* any history of ophthalmic surgeries
* evidence of serious ocular or brain pathologies affecting visual acuity (VA)
* clinically active inflammation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Visual Acuity based on The Early Treatment Diabetic Retinopathy Study protocol | day one
  Examination for visual performance in 3 trials: reference (with lens for distance correction); stenopeic (distance correction with a pinhole ϕ=1,25 mm) and Light Sword Lens (distance correction with a Light Sword Lens). In each trial, visual acuity assessment in 7 tasks for defocus from 0.2D to 3.0D.
  The degree of homogeneity through defocus was determined. Reference and stenopeic trials were compared to Light Sword Lens results.
  Statistical analysis: Friedman analysis of variance, Nemenyi post-hoc, Wilcoxon tests , p-value < 0.05 is considered significant.
Contrast sensitivity based on Pelli-Robson method | day one
  Contrast sensitivity assessment in 2 tasks for defocus 0.3D and 2.5D The degree of homogeneity through defocus was determined. Reference and stenopeic trials were compared to Light Sword Lens results.
  Statistical analysis: Friedman analysis of variance, Nemenyi post-hoc, Wilcoxon tests , p-value < 0.05 is considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Petelczyc, PhD, Study Director — Warsaw University of Technology

IPD SHARING:
Plan to Share IPD: Yes
data will be supplemented to published outcomes
Supporting Information: Study Protocol
Time Frame: data will be supplemented to published outcomes

REFERENCES:
- [Background] Kakarenko K, Ducin I, Grabowiecki K, Jaroszewicz Z, Kolodziejczyk A, Mira-Agudelo A, Petelczyc K, Skladowska A, Sypek M. Assessment of imaging with extended depth-of-field by means of the light sword lens in terms of visual acuity scale. Biomed Opt Express. 2015 Apr 16;6(5):1738-48. doi: 10.1364/BOE.6.001738. eCollection 2015 May 1. PMID 26137376
- [Background] Mira-Agudelo A, Torres-Sepulveda W, Barrera JF, Henao R, Blocki N, Petelczyc K, Kolodziejczyk A. Compensation of Presbyopia With the Light Sword Lens. Invest Ophthalmol Vis Sci. 2016 Dec 1;57(15):6870-6877. doi: 10.1167/iovs.16-19409. PMID 28002561